CLINICAL TRIAL: NCT01351116
Title: A Phase III, Multi-centre, Randomized Trial to Evaluate the Symptomatic and Quality of Life Improvements in Lung Cancer Patients Receiving External Beam Radiation With or Without High Dose Rate Intraluminal Brachytherapy
Brief Title: A Trial to Evaluate the Improvement in Lung Cancer Patients Receiving Radiation With or Without Brachytherapy
Acronym: BRACHY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2011-BRACHY
Record Dates: First submitted 2011-05-02; First posted 2011-05-10 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: brachytherapy; external beam radiation; high dose rate intraluminal brachytherapy; lung cancer; quality of life; radiation treatment; bronchus
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EBR plus HDRIB (Experimental): External Beam Radiation (EBR) plus High Dose Rate Intraluminal Brachytherapy (HDRIB)
  Interventions: Radiation: EBR plus HDRIB
- EBR (Active Comparator): External Beam Radiation (EBR)
  Interventions: Radiation: EBR

INTERVENTIONS:
Radiation: EBR plus HDRIB — EBR of 20 Gy in 5 daily fractions over one week plus HDRIB of 14 Gy in 2 fractions over two weeks
  Arms: EBR plus HDRIB
Radiation: EBR — EBR of 20 Gy in 5 daily fractions over one week
  Arms: EBR

SUMMARY:
A trial to improve the quality of life of patients with advanced non-small cell lung cancer (NSCLC) by evaluating the symptomatic improvements in lung cancer patients receiving external radiation with or without high dose internal radiation.

DETAILED DESCRIPTION:
In patients with advanced NSCLC to compare the added benefit of High Dose Rate Intraluminal Brachytherapy (HDRIB) with External Beam Radiation (EBR). Benefit will be assessed by measuring the proportion of patients who achieve symptomatic improvement in lung cancer symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic proof of non-small cell lung cancer (NSCLC)
* Stages III, IV or recurrent disease
* Documented endobronchial luminal disease by either endoscopy or CT-imaging
* Candidate for palliative thoracic radiation therapy because of cough, shortness of breath or hemoptysis

Exclusion Criteria:

* Age less than 18 years of age
* Uncontrolled or symptomatic brain metastases
* Anticipated survival of less than 3 months
* Systemic therapy planned to begin within 6 weeks following randomization
* Systemic therapy within 4 weeks of planned study randomization
* Any prior radiotherapy involving the lungs
* Cardiac arrest or myocardial infarction within 6 months prior to study randomization
* Inability to receive sedation or undergo invasive procedures due to severe chronic obstructive pulmonary disease (COPD), bleeding disorders, or other medical conditions which will preclude the use of HDRIB
* Pregnancy, lactation, or failure to use dual-method contraception in pre-menopausal women
* Unwillingness or inability (e.g. incompetence, severe psychiatric disorders) to complete informed consent and the baseline QoL assessments required for the trial
* Having received an investigational agent within one month of study randomization
* Inability to attend regular follow-up evaluations due to psychiatric or addictive disorder or geographic inaccessibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-10; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
For each subject, a lung cancer-related symptomatic improvement at 6 weeks post randomization, defined as a 10-point improvement on a 100 point scale from the summary question of lung cancer symptoms | 6 weeks from randomization

SECONDARY OUTCOMES:
Improvement in each lung cancer symptom as measured by the Lung Cancer Symptom Scale (LCSS) as defined by a 10-point improvement for cough, shortness of breath, hemoptysis and pain on the LCSS at 6 weeks post randomization | 6 weeks post randomization
Improvement in each lung cancer symptom and overall symptoms at any time after randomization | at 3, 6, 12, 18, 26, 34, 42 and 50 weeks post-randomization
A Quality of Life (QOL) improvement as measured be overall score of the LCSS, at each scheduled assessment point following randomization (Weeks 3, 6, 12, 26, 34, 42 and 50) | Weeks 3, 6, 12, 18, 26, 34, 42 and 50
Symptomatic progression-free survival (SPFS), defined as the time from randomization until death, use of chemotherapy, or the first post-randomization score on LCSS #7 which is 10 points or greater than the baseline score, or scored at 100. | From date of randomization until the date of first documented use of chemotherapy, or progression whichever came first, assessed up to 48 months
Overall survival, calculated from the date of randomization to the date of death | From date of randomization until the date of death from any cause assessed up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Ranjan Sur, Principal Investigator — Juravinski Cancer Centre
Locations (8):
- Canada (8):
  - Abbotsford Centre - BC Cancer Agency, Abbotsford, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Centre, London, Ontario
  - UHN-Princess Margaret Cancer Centre, Toronto, Ontario
  - Windsor Regional Hospital Cancer Centre, Windsor, Ontario
  - CHUQ - L'Hôtel-Dieu de Québec, Québec, Quebec